CLINICAL TRIAL: NCT02946957
Title: Efficacy of Scalable CBT for Insomnia in Older Adults With Osteoarthritis Pain
Brief Title: OsteoArthritis and Therapy for Sleep
Acronym: OATS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Michael Vitiello, Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52176
Record Dates: First submitted 2016-10-19; First posted 2016-10-27 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Insomnia Related to Osteoarthritis Pain
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Cognitive Behavioral Therapy for Insomnia is delivered by trained sleep therapists in six telephone sessions.
  Interventions: Behavioral: Cognitive Behavior Therapy for Insomnia
- Education Control (Active Comparator): Education Only Control is delivered by trained sleep therapists in six telephone sessions.
  Interventions: Behavioral: Education Only Control

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy for Insomnia — Six telephone sessions that last 20-30 minutes presenting cognitive behavioral therapy for insomnia.
  Other Names: CBT-I
  Arms: Cognitive Behavioral Therapy
Behavioral: Education Only Control — Six telephone sessions that last 20-30 minutes presenting sleep and osteoarthritis education.
  Other Names: EOC
  Arms: Education Control

SUMMARY:
Osteoarthritis (OA) pain affects 50 percent of older adults, more than half of whom also experience significant sleep disturbance. This randomized trial will determine whether a telephone-based cognitive behavioral treatment targeting insomnia in older adults with chronic severe OA-related insomnia and pain results in substantially greater reductions in insomnia severity and in related improvements in pain, fatigue, mood, quality of life and healthcare costs compared to telephone-delivered education (attention control) about insomnia. The trial will test an intervention that if demonstrated to have long term efficacy is scalable and has the potential for wide-scale deployment in healthcare systems.

DETAILED DESCRIPTION:
Twenty-five percent of older adults experience significant osteoarthritis (OA)-related comorbid sleep disturbance. Insomnia is associated with substantial negative effects on function, mood, and medical resource utilization. Cognitive behavioral therapy for insomnia (CBT-I) is evidence based and has been shown to be efficacious in populations with a variety of comorbid conditions including OA-related chronic pain. However, in-person CBT interventions are unlikely to be widely deployable in healthcare systems. Telephone delivery has the advantage of giving patients access to personalized, efficacious CBT-I interventions from home, increasing generalizability, and outreach to minority, rural, and other underserved populations. Older (60+ yrs) primary care patients across Washington State will be screened for severe persistent OA-related insomnia and pain. Two hundred and seventy patients will be randomized to either CBT-I or an education only attention control (EOC). Each treatment will consist of six 20-30 minute telephone-based sessions over an eight week period. Pre-treatment, post-treatment (2 months and 12 month) assessments will include measures of sleep, pain, fatigue, mood, and quality of life. A cost effectiveness evaluation of the intervention will also be conducted. The proposed research will determine if telephone CBT-I improves OA insomnia and associated outcomes in a state-wide primary care population of older adults, and inform policy decisions about widespread dissemination of telephone CBT-I in this and related patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Age 60+ with one or more health care visits for OA in the prior 3 years
* Score of ≥6 on 4-item ISI at first screening and ≥11 on full ISI at second screening
* Score of ≥9 on two items from the Brief Pain Inventory (BPI) asking about average pain intensity in the past 2 weeks (0-10 scale) and activity interference due to pain (0-10 scale) at first and second screening

Exclusion Criteria:

* Not continuously enrolled at Group Health Cooperative for at least one year
* Prior diagnosis of a primary sleep disorder: sleep apnea with an AHI/RDI score of 15+ or current use of a CPAP machine; periodic leg movement disorder; restless leg syndrome; sleep-wake cycle disturbance; or rapid eye movement behavior disorder
* Diagnosis in the medical record of: rheumatoid arthritis, terminal disease, being considered for major surgery, active chemotherapy or radiation for cancer, or inpatient treatment for congestive heart failure within the previous 6 months
* Diagnosis of dementia, use of acetylcholinesterase inhibitor and/or memantine for cognitive impairment, or cognitive impairment (>6 on the Short Orientation-Memory-Concentration Test)
* Hearing or speech impairment sufficient to preclude participation in a telephone intervention

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2016-10; Primary Completion 2019-12 (Actual); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 12 months post baseline
  A 7-item questionnaire that is a global measure of perceived insomnia severity. Items use a 5-point scale for total scores of 0-28, with >15 considered moderate severity.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | 2 months post baseline
  A 7-item questionnaire that is a global measure of perceived insomnia severity.Items use a 5-point scale for total scores of 0-28, with >15 considered moderate severity.
Pittsburgh Sleep Quality Index (PSQI) | 2 months post baseline
  Self-rating of overall sleep quality and disturbances using 7 sleep. components. PSQI global >5 is highly sensitive and specific for distinguishing good and poor sleepers.
Pittsburgh Sleep Quality Index (PSQI) | 12 months post baseline
  Self-rating of overall sleep quality and disturbances using 7 sleep components. PSQI global >5 is highly sensitive and specific for distinguishing good and poor sleepers.
Brief Pain Inventory-short form (BPI-sf) | 2 months post baseline
  A questionnaire to assess pain intensity and interference with activities. The BPI-sf rates pain intensity (4 items) and interference (7 items) from 0 to 10 and is validated for use in clinical trials with OA pain patients.
Brief Pain Inventory-short form (BPI-sf) | 12 months post baseline
  A questionnaire to assess pain intensity and interference with activities. The BPI-sf rates pain intensity (4 items) and interference (7 items) from 0 to 10 and is validated for use in clinical trials with OA pain patients.
Flinders Fatigue Scale (FFS) | 2 months post baseline
  A 7-item self-report questionnaire to measure fatigue level in a variety of situations.
Flinders Fatigue Scale (FFS) | 12 months post baseline
  A 7-item self-report questionnaire to measure fatigue level in a variety of situations.
Patient Health Questionnaire (PHQ-8) | 2 months post baseline
  4-point scale rates frequency of occurrence of 8 depressive symptoms.
Patient Health Questionnaire (PHQ-8) | 12 months post baseline
  4-point scale rates frequency of occurrence of 8 depressive symptoms.
Sleep Hygiene Index (SHI) | 2 months post baseline
  A 13-item scale that rates how often participants engage in specific sleep hygiene related behaviors, including continued adherence to CBT-I recommendations over time.
Sleep Hygiene Index (SHI) | 12 months post baseline
  A 13-item scale that rates how often participants engage in specific sleep hygiene related behaviors, including continued adherence to CBT-I recommendations over time.
EuroQoL 5D (EQ-5D) | 2 months post baseline
  Rates health status on five dimensions and overall health status from 0 to 100. The most widely used measure in clinical trials assessing general quality of life of OA patients.
EuroQoL 5D (EQ-5D) | 12 months post baseline
  Rates health status on five dimensions and overall health status from 0 to 100. The most widely used measure in clinical trials assessing general quality of life of OA patients.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 2 months post baseline
  A 24-item questionnaire rating pain, stiffness, and physical functioning in everyday activities. It is the most widely used condition-specific quality of life measure for arthritis cost-effectiveness studies.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 12 months post baseline
  A 24-item questionnaire rating pain, stiffness, and physical functioning in everyday activities. It is the most widely used condition-specific quality of life measure for arthritis cost-effectiveness studies.
Use of sleep and pain medications | Baseline through 24 months
  NSAID, analgesic, sedative, and anti-depressant medication use.
Outpatient visits | Baseline through 24 months
  The number of visits for OA, for sleep problems, and for visits irrespective of associated diagnosis.
Health care costs | Baseline through 24 months
  The Group Health cost database will be used to estimate costs (from study entry to 24 months post enrollment) of ambulatory healthcare for all conditions, arthritis and sleep problems, and inpatient care.

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Vitiello, PhD, Principal Investigator — University of Washington; Susan M McCurry, PhD, Principal Investigator — University of Washington; Michael Von Korff, ScD, Principal Investigator — University of Washington; Kai Yeung, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vitiello MV, Zhu W, Von Korff M, Wellman R, Morin CM, Yeung K, McCurry SM. Long-term improvements in sleep, pain, depression, and fatigue in older adults with comorbid osteoarthritis pain and insomnia. Sleep. 2022 Feb 14;45(2):zsab231. doi: 10.1093/sleep/zsab231. PMID 34516646
- [Derived] Thakral M, Von Korff M, McCurry SM, Morin CM, Vitiello MV. ISI-3: evaluation of a brief screening tool for insomnia. Sleep Med. 2021 Jun;82:104-109. doi: 10.1016/j.sleep.2020.08.027. Epub 2020 Aug 27. PMID 33910159
- [Derived] McCurry SM, Zhu W, Von Korff M, Wellman R, Morin CM, Thakral M, Yeung K, Vitiello MV. Effect of Telephone Cognitive Behavioral Therapy for Insomnia in Older Adults With Osteoarthritis Pain: A Randomized Clinical Trial. JAMA Intern Med. 2021 Apr 1;181(4):530-538. doi: 10.1001/jamainternmed.2020.9049. PMID 33616613
- [Derived] McCurry SM, Von Korff M, Morin CM, Cunningham A, Pike KC, Thakral M, Wellman R, Yeung K, Zhu W, Vitiello MV. Telephone interventions for co-morbid insomnia and osteoarthritis pain: The OsteoArthritis and Therapy for Sleep (OATS) randomized trial design. Contemp Clin Trials. 2019 Dec;87:105851. doi: 10.1016/j.cct.2019.105851. Epub 2019 Oct 13. PMID 31614214